CLINICAL TRIAL: NCT00320658
Title: Phase 1 Study of the Safety and Immunogenicity of MSP1 42-C1/Alhydrogel With and Without CPG 7909, an Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria
Brief Title: Safety of and Immune Response to a Malaria Vaccine (MSP1 42-C1) With or Without CPG 7909 Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 212; NIH Protocol Number 05-I-0240; WIRB Protocol Number 20051029; NCT00342420 (obsolete NCT alias)
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Malaria
Keywords: Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — ProMune

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): 3 vaccinations with a dose of 40 mcg MSP1 42-C1/Alhydrogel given into the deltoid muscle of either arm. Each vaccination will be given 1 month apart. This arm will enroll concurrently with Arm B.
  Interventions: Biological: MSP1 42-C1/Alhydrogel
- B (Experimental): 3 vaccinations with a dose of 40 mcg MSP1 42-C1/Alhydrogel and CPG7909 given into the deltoid muscle of either arm. Each vaccination will be given 1 month apart. This arm will enroll concurrently with Arm A.
  Interventions: Biological: MSP1 42-C1/Alhydrogel; Biological: CPG 7909
- C (Experimental): 3 vaccinations with a dose of 160 mcg MSP1 42-C1/Alhydrogel given into the deltoid muscle of either arm. Each vaccination will be given 1 month apart. This arm will enroll concurrently with Arm D after review of the results from Arms A and B.
  Interventions: Biological: MSP1 42-C1/Alhydrogel
- D (Experimental): 3 vaccinations with a dose of 160 mcg MSP1 42-C1/Alhydrogel and CPG7909 given into the deltoid muscle of either arm. Each vaccination will be given 1 month apart. This arm will enroll concurrently with Arm C after review of the results from Arms A and B.
  Interventions: Biological: MSP1 42-C1/Alhydrogel; Biological: CPG 7909

INTERVENTIONS:
Biological: MSP1 42-C1/Alhydrogel — Recombinant MSP1 42-C1/Alhydrogel vaccine (one of two doses)
Biological: CPG 7909 — Adjuvant
  Arms: B; D

SUMMARY:
The purpose of this study is to determine the safety of and immune response to a preventive malaria vaccine, MSP1 42-C1/Alhydrogel, in healthy adults. This study will also compare responses to two different doses of the malaria vaccine given with or without the adjuvant CPG 7909.

DETAILED DESCRIPTION:
In 2002, the World Health Organization reported a worldwide malaria incidence of approximately 300 million clinical cases annually, with approximately 1 million deaths attributed to malaria alone or in combination with other diseases. The parasite Plasmodium falciparum is responsible for the majority of these infections and deaths. During P. falciparum infection, liver cells are invaded by the parasite and asexual multiplication occurs. The liver cells burst, and tens of thousands of infectious particles called merozoites are released. A multiprotein complex on the surface of a merozoite is necessary for the merozoite to infect a blood cell. MSP1 42-C1 is a malaria vaccine that mimics MSP1 42, a protein in the multiprotein complex. By introducing this "decoy" form of MSP1 42, infection of additional blood cells may be blocked. The adjuvant CPG 7909 is known to elicit cell-mediated immunity, the arm of the immune system that defends the body against intracellular pathogens such as P. falciparum. This study will evaluate the safety and immunogenicity of MSP1 42-C1/Alhydrogel at two different doses in healthy adults. The vaccine will be given either alone or with CPG 7909.

This study will last at least 34 weeks. Participants will be randomly assigned to one of four groups:

* Group A participants will receive three injections of the lower dose of MSP1 42-C1/Alhydrogel.
* Group B participants will receive three injections of the lower dose of MSP1 42-C1/Alhydrogel and CPG 7909.
* Group C participants will receive three injections of the higher dose of MSP1 42-C1/Alhydrogel.
* Group D participants will receive three injections of the higher dose of MSP1 42-C1/Alhydrogel and CPG 7909.

Enrollment into Groups C and D will begin only after safety review of all participants in Groups A and B. All participants will receive their assigned injections at study entry, Week 4, and Week 8, and will be asked to return to the clinic the day after each vaccination for clinical evaluation. Participants will be asked to keep a diary for 6 days after each vaccination, taking note of their body temperatures and any side effects they experience. There will be a total of 18 study visits over 34 weeks. A clinical evaluation will occur at each visit. Blood collection, vital signs measurement, and urine collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Willing to be followed for the duration of the study
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may affect the ability of the volunteer to understand and cooperate with the study
* Liver disease (ALT greater than upper limit of normal [ULN])
* Kidney disease (serum creatinine greater than ULN)
* Hematologic disease (absolute neutrophil count of less than 1,500 cells/mm3; hemoglobin less than lower limit of normal, by sex; OR platelet count less than 140,000 mm3)
* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Participation in another investigational vaccine or drug trial within 30 days of study entry or while this study is ongoing
* Active drug or alcohol abuse causing medical, occupational, or family problems during the 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* HIV-1 infected
* Hepatitis C virus infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Blood products within 6 months prior to study entry
* Absence of spleen
* Previously received an investigational malaria vaccine
* Received antimalarial prophylaxis during the 12 months prior to study entry
* Received chloroquine or other aminoquinolines within 12 weeks of study entry
* Prior malaria infection
* Known allergy to nickel
* Pre-existing autoimmune or antibody-mediated disease. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, social, or occupational condition or other responsibility that, in the opinion of the investigator, would interfere with the study
* Other condition that, in the opinion of the investigator, would affect the volunteer's participation in the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events, as classified by both intensity and severity through active and passive surveillance | Throughout study
Anti-MSP1 42 antibody concentration as measured by ELISA | At Day 70

SECONDARY OUTCOMES:
To demonstrate that the addition of CPG 7909 improves the specific immune responses to MSP142-FVO and MSP142-3D7, as compared to MSP142-C1/Alhydrogel | At Day 70
To determine the dose of MSP142-C1/Alhydrogel + CPG 7909 that generates the highest serum antibody levels of MSP142-FVO and MSP142-3D7 | At Day 70

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins University, Bloomberg School of Public Health, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Boutlis CS, Riley EM, Anstey NM, de Souza JB. Glycosylphosphatidylinositols in malaria pathogenesis and immunity: potential for therapeutic inhibition and vaccination. Curr Top Microbiol Immunol. 2005;297:145-85. doi: 10.1007/3-540-29967-x_5. PMID 16265905
- [Background] Hill AV. Pre-erythrocytic malaria vaccines: towards greater efficacy. Nat Rev Immunol. 2006 Jan;6(1):21-32. doi: 10.1038/nri1746. PMID 16493425
- [Background] Reed ZH, Friede M, Kieny MP. Malaria vaccine development: progress and challenges. Curr Mol Med. 2006 Mar;6(2):231-45. doi: 10.2174/156652406776055195. PMID 16515513
- [Background] Saul A, Lawrence G, Smillie A, Rzepczyk CM, Reed C, Taylor D, Anderson K, Stowers A, Kemp R, Allworth A, Anders RF, Brown GV, Pye D, Schoofs P, Irving DO, Dyer SL, Woodrow GC, Briggs WR, Reber R, Sturchler D. Human phase I vaccine trials of 3 recombinant asexual stage malaria antigens with Montanide ISA720 adjuvant. Vaccine. 1999 Aug 6;17(23-24):3145-59. doi: 10.1016/s0264-410x(99)00175-9. PMID 10462251
- [Derived] Ellis RD, Martin LB, Shaffer D, Long CA, Miura K, Fay MP, Narum DL, Zhu D, Mullen GE, Mahanty S, Miller LH, Durbin AP. Phase 1 trial of the Plasmodium falciparum blood stage vaccine MSP1(42)-C1/Alhydrogel with and without CPG 7909 in malaria naive adults. PLoS One. 2010 Jan 22;5(1):e8787. doi: 10.1371/journal.pone.0008787. PMID 20107498